CLINICAL TRIAL: NCT01836120
Title: A Study of Raltitrexed Plus Docetaxel Versus Docetaxel as Second-line Chemotherapy in Subjects With Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hebei Tumor Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HBTH103
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Gastric Cancer
Keywords: second-line chemotherapy; Raltitrexed
MeSH Terms: conditions — Stomach Neoplasms | interventions — raltitrexed; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raltitrexed plus Docetaxel (Experimental)
  Interventions: Drug: Raltitrexed plus Docetaxel
- Docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Raltitrexed plus Docetaxel — Raltitrexed plus Docetaxel (Raltitrexed 3mg/m2 d
  1; Docetaxel 75mg/m2 d1, every 3 weeks, 4-6 cycles)
  Arms: Raltitrexed plus Docetaxel
Drug: Docetaxel — Docetaxel (Docetaxel 75mg/m2 d1, every 3weeks,4-6 cycles)
  Arms: Docetaxel

SUMMARY:
A study of Raltitrexed plus Docetaxel versus Docetaxel as second-line chemotherapy in subjects with Gastric Cancer.The purpose of this study is to compare the activity of Raltitrexed plus Docetaxel versus Docetaxel as second-line chemotherapy in subjects with gastric carcinoma by estimating progression free survival (PFS) in each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-2;
3. Histologically or cytologically confirmed gastric cancer;
4. The first-line chemotherapy failure (required containing 5-fluorouracil)
5. At least have one measurable disease(according to RECIST, Response Evaluation Criteria in Solid Tumors )
6. Life expectancy of at least 3 months;

Exclusion Criteria:

1. Received any prior treatment including Raltitrexed;
2. Active or uncontrolled infection;
3. Concurrent treatment with an investigational agent or participation in another therapeutic clinical trial;
4. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 1 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 1 year
Overall Survival (OS) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Tumor Hospital, Shijiazhuang, Hebei, China